CLINICAL TRIAL: NCT05967884
Title: A Randomized Phase II Window of Opportunity Clinical Trial of IL-4 +/- PD-1 Inhibition in Early-stage ER+ HER2- Breast Cancer
Brief Title: PD-1 +/- IL-4 Inhibition in ER+ Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Ontario Institute for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMS 05-2023
Record Dates: First submitted 2023-07-12; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer
Keywords: Window of Opportunity Clinical Trials; cemiplimab; dupilumab
MeSH Terms: conditions — Breast Neoplasms | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Cemiplimab (Active Comparator): Arm A: Cemiplimab (n=10), 350mg IV x 1 dose administered prior to surgery.
  Interventions: Drug: Arm A: Cemiplimab, Arm B: Cemiplimab + Dupilumab
- Arm B: Cemiplimab + Dupilumab (Experimental): Arm B: Cemiplimab + Dupilumab (n=10), Cemiplimab 350mg IV x 1 dose + Dupilumab 600 mg SC x 1 dose administered prior to surgery.
  Interventions: Drug: Arm A: Cemiplimab, Arm B: Cemiplimab + Dupilumab

INTERVENTIONS:
Drug: Arm A: Cemiplimab, Arm B: Cemiplimab + Dupilumab — Arm A: Cemiplimab: 350mg IV x 1 dose administered prior to surgery Arm B: Cemiplimab + Dupilumab: Cemiplimab 350mg IV x 1 dose + Dupilumab 600 mg SC x 1 dose administered prior to surgery

SUMMARY:
This proposal is for a Window of Opportunity (WOO) clinical trial using a novel combination of two Health Canada approved agents, cemiplimab (Libtayo) and dupilumab (Dupixent), for off label use in early-stage estrogen receptor positive (ER+) breast cancer.

DETAILED DESCRIPTION:
This is a phase II, open-label, randomized window of opportunity trial evaluating the immunologic effects within the tumour, microenvironment, and host blood of patients treated with either

* Arm A: Cemiplimab (n=10)
* Arm B: Cemiplimab + Dupilumab (n=10) administered prior to surgery. Randomization will be at 1:1 ratio in patients newly diagnosed with primary operable ER+* HER2- invasive breast cancer awaiting surgery in the next 4-6 weeks who are not planned for neoadjuvant therapy.

Primary Hypothesis: In ER+ breast cancer, blockade of IL-4 signalling using dupilumab enhances anti-tumor immunity (through reduced Th2 skewing) when used in combination with PD-1 inhibitors (Cemiplimab) compared to PD-1 inhibition alone in ER+ breast cancer

Primary Objective:

• To determine whether addition of dupilumab to cemiplimab reduces TH2 skewing of the tumor, tumor microenvironment (TME) and blood in patients with ER+ breast cancer

Secondary Objectives:

* To evaluate dynamic changes in immune cell populations as measured by in situ proteomics
* To characterize the safety of a short-term duration of the combination of dupilumab with cemiplimab in patients with ER+ breast cancer awaiting surgery

Exploratory Objective:

• To test the effect of tumor PD-1 gene expression and its effect on the immune response in treated and untreated patients

This is a window of opportunity trial which will require administration of cemiplimab or combination of cemiplimab + dupilumab prior to surgery. Surgery will be a minimum of 96 hours to 2 weeks after the cemiplimab. Patient follow-up after surgery will be for a period of 30 days post-surgery.

Target: 20 patients (10 in Arm A and 10 in Arm B). Accounting for screen failures and withdrawals (20%), 24 patients will be accrued.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with newly diagnosed histologically confirmed primary invasive breast cancer currently not undergoing any treatment while awaiting surgery.
2. Invasive ductal or lobular carcinoma, invasive carcinoma Not Otherwise Specified (NOS)
3. ER+ breast cancer (1-10%*) of any size. ER positive tumor defined ≥1% positively staining cells by immunohistochemistry, according to the current American Society of Clinical Oncology (ASCO) / College of American Pathologists (CAP) guidelines.
4. The participant is eligible for surgery within the next 4-6 weeks.
5. HER2/neu must be negative by immunohistochemistry (IHC) defined as IHC 0 or 1+ or fluorescence in situ hybridization (FISH) or other ISH methods with a ratio of < 2 according to current ASCO (American Society of Clinical Oncology)/CAP guidelines.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
7. Age ≥18 years.
8. The participant (or legally acceptable representative if applicable) is able to provide written informed consent for the study.

Exclusion Criteria:

1. Known or suspected breast cancer metastasized to distant organ (lung, liver, bone, brain, abdomen)
2. Prior therapy with any chemotherapy or endocrine for breast cancer or other cancers within last 3 months
3. Pre-dominant histology other than invasive ductal or lobular carcinoma or invasive carcinoma NOS.
4. Patients with an active infection or an absolute neutrophil count < 1.5 x 10^9/L.

6. Patients with pre-existing renal impairment, Creatinine clearance calculated by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation of less than 50 mL/min/1.73m2.

7. Known or current history of pneumonitis or interstitial lung disease (e.g., idiopathic pulmonary fibrosis) or pneumonia in past month 8. Has known HIV or active Hepatitis B (e.g., HBV detected by PCR, presence of HBsAg surface antigen and/or Anti-HBc core antigen) or active Hepatitis C (e.g., HCV RNA [qualitative] is detected). Presence of Anti-HBs alone suggesting immunity to Hepatis B is eligible.

9. Any serious known immediate or delayed hypersensitivity reaction(s) to dupilumab and or cemiplimab.

10. Concurrent medical condition requiring the use of systemic immunosuppressive medications, or systemic corticosteroids at doses of greater than 10 mg Prednisone-equivalent. Topical steroids and other localized corticosteroids are permitted. Patients who have received acute, low-dose, systemic immunosuppressant medications equivalent to ≤ 10mg of prednisone within the 7 days prior to study entry (small dose of dexamethasone for nausea, short course for upper respiratory tract infection etc.) may be enrolled in the study. Use of steroids as prophylactic treatment for subjects with contrast allergies to diagnostic imaging contrast dyes will be permitted.

11. Concurrent use or planned use of any forbidden medications within 4 weeks prior to study drug administration, which include chemotherapy, immunotherapy (tumor vaccine, cytokine, or growth factor given to control cancers), other biologic therapy, investigational therapy, or hormonal therapy.

12. Confirmed pregnancy (by pregnancy test) if patient is of childbearing age or breast feeding.

13. Subjects with signs/symptoms suggestive of COVID-19 and confirmed positive COVID-19 test.

14. Eastern Cooperative Oncology Group (ECOG) performance status ≥3 (see Appendix) 15. Any underlying medical condition that, in the Principal Investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity determination or adverse events, or renders the patient ineligible to be on study.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-04 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Immune Cell Population Analysis | up to 6 months
  The % change in various immune cell populations (CD3, CD8, macrophages and DC cells) in the tumor and microenvironment, Defined as the post-treatment value / pre-treatment value * 100%

SECONDARY OUTCOMES:
Study Participant Assessment of Adverse Effects | up to 6 months
  Number of participants with treatment-related adverse effects of patients treated with short term cemiplimab + dupilumab, using NCI-CTCAE

OTHER OUTCOMES:
PD-1 Gene Expression | up to 6 months
  PD-1 Gene expression analysis in pre treatment tissue samples expression and its effect on the immune response in treated and untreated patients

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - The Ottawa Hospital Research Institute and Cancer Center, Ottawa, Ontario
  - Ontario Institute for Cancer Research, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
undecided